CLINICAL TRIAL: NCT00914862
Title: A Comparative Single Dose Pharmacokinetic and Safety Study of 4 mg or 8 mg Ramelteon in Adolescents With Insomnia Characterized by Difficulty With Sleep Onset, Children With Insomnia Associated With ADHD, and Healthy Adults.
Brief Title: Pharmacokinetic and Safety of Ramelteon Between Adolescents With Insomnia and Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TAK-375_110; U1111-1112-5188 (Registry Identifier: WHO)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-03

CONDITIONS: Insomnia
Keywords: Sleep Initiation and Maintenance Disorders; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Children Ramelteon 4 mg (Experimental): Children 6 to 11 years of age who had insomnia associated with ADHD received a single 4 mg oral dose of ramelteon.
  Interventions: Drug: Ramelteon
- Children Ramelteon 8 mg (Experimental): Children 6 to 11 years of age who had insomnia associated with ADHD received a single oral 8 mg dose of ramelteon.
  Interventions: Drug: Ramelteon
- Adolescents Ramelteon 4 mg (Experimental): Adolescents 12 to 17 years of age with insomnia received a single oral dose of 4 mg ramelteon.
  Interventions: Drug: Ramelteon
- Adolescents Ramelteon 8 mg (Experimental): Adolescents 12 to 17 years of age with insomnia received a single oral dose of 8 mg ramelteon.
  Interventions: Drug: Ramelteon
- Healthy Adult Ramelteon 8 mg (Active Comparator): Healthy adults (18 to 50 years old) received a single oral dose of 8 mg ramelteon.
  Interventions: Drug: Ramelteon

INTERVENTIONS:
Drug: Ramelteon — Ramelteon tablets, orally for one day only.
  Other Names: TAK-375; Rozerem

SUMMARY:
The purpose of this study is to determine the pharmacokinetic profile, safety, and tolerability of ramelteon in adolescents with insomnia, children with Attention Deficit Hyperactivity Disorder (ADHD) associated with insomnia and gender- and race-matched healthy adults.

DETAILED DESCRIPTION:
Ramelteon is a treatment for insomnia approved for use in the United States (US) in July 2005 and in the Philippines and Indonesia in 2008. It is currently under development in the European Union (EU) and Japan. Ramelteon is marketed in the US as ROZEREM® for the treatment of insomnia characterized by difficulty with sleep onset in patients over 18 years of age.

In adolescents, the form of sleep onset and/or sleep maintenance insomnia, defined as psychophysiologic insomnia, is similar to adults, and more appropriate for treatment with pharmacological intervention when compared to insomnia in children younger than 12 years of age. In psychophysiologic insomnia, the individual develops conditioned anxiety around difficulty falling or staying asleep, which leads to heightened physiologic and emotional arousal and further compromises the ability to sleep. In children over the age of 12, insomnia is more likely to be persistent and have identifiable consequences. In addition, there is less variability in normative sleep data for this age group than in younger children.

Sleep disturbances are also common in children. Specifically, insomnia associated with ADHD in children is very common with a reported prevalence of 28% in medication-free children with ADHD.

This study is to characterize the pharmacokinetics (PK) and safety profile of a 4 or 8 mg dose of ramelteon in adolescents who are between 12 to 17 years of age (prior to the 18th birthday) with insomnia characterized by difficulty with sleep initiation, and in pediatrics who are between 6 to 11 years of age who have insomnia associated with ADHD. These profiles will be compared with those of healthy adults aged 18 to 50 years who are matched by race and gender receiving an 8 mg dose of ramelteon. This open-label study is designed in accordance with the recommendations of the FDA and ICH guidances for pediatric PK studies.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for adolescent and pediatric participants only:

* Is male or female between 12 and 17 years of age (less than 18 years of age on Day 1) with complaints of insomnia characterized by difficulty with sleep initiation OR a male or female between 6 to 11 years of age (less than 12 years of age on Day 1) with complaints of insomnia characterized by difficulty with sleep initiation associated with ADHD.
* Has a body mass index within the 5th to 95th percentile of the appropriate body mass index designated charts based on stature-for-age and weight-for-age and by gender.
* In the age group of 12 to 17 years, has a history of primary insomnia characterized by difficulty initiating sleep as defined by the Pharmacologic Management of Insomnia in Children and Adolescents: Consensus Statement OR in the age group of 6 to 11 years, has a history of insomnia characterized by difficulty with sleep initiation (as defined by the Pharmacologic Management of Insomnia in Children and Adolescents: Consensus Statement associated with ADHD).
* There is agreement in the participant's parent or caregiver's opinion with the following:

  * The complaint involves significant difficulty in initiating sleep
  * The sleep disturbance does not occur exclusively during the course of narcolepsy, breathing-related sleep disorder, circadian rhythm sleep disorder, or parasomnia.
  * The disturbance does not occur exclusively during the course of another mental disorder (eg, Major Depressive Disorder, Generalized Anxiety Disorder, and Delirium).
  * The disturbance is not due to the direct physiological effects of a substance (eg, a drug of abuse, a medication) or a general medical condition.
* Based on sleep history, reports a subjective sleep latency greater than or equal to 45 minutes for at least 1 month.
* If taking concomitant medications, he/she has been on a stable dose or regimen of his/her medication for at least 30 days prior to Screening.

Inclusion criteria for gender- and race-matched adult participants only:

* Weighs at least 50 kg (110 pounds) and has a Screening body mass index between 18 and 30 kg/m^2, inclusive.

Inclusion criteria for all participants:

* A female of childbearing potential (defined as females aged ≥12 years old and younger girls who, at the discretion of the investigator, are deemed to be of reproductive potential) and males who are sexually active agree to routinely use adequate contraception from Screening throughout the duration of the study and through 30 days following the last dose of study medication.
* Must have a negative urine test result for selected substances of abuse (including alcohol) at Screening and Day 1.
* Has clinical laboratory results (including clinical chemistry, hematology, and complete urinalysis [fasted] within the reference range for the testing laboratory unless the results are deemed not clinically meaningful by the investigator or sponsor.
* Has a negative test result for hepatitis B surface antigen and hepatitis C virus antibody, and no known history of human immunodeficiency virus.

Exclusion Criteria:

* Is participating in another investigational study or has taken an investigational drug within 30 days (or 5 half-lives, whichever period is longer) prior to study Screening.
* Has received ramelteon within 30 days of Screening.
* Is a study site employee, or is an immediate family member (ie, spouse, parent, child, sibling) of a study site employee, involved in conduct of this study.
* Has abnormal hematological parameters of hemoglobin and/or hematocrit (if these exceed +/- 2 points of the normal range for the age and sex appropriate values), or erythrocytes at Screening.
* Has a known hypersensitivity to ramelteon or related compounds including melatonin.
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as consumption of more than 4 alcoholic drinks per day) within 1 year prior to study Day 1.
* Has had an acute, clinically significant illness within 30 days prior to Screening.
* Has autistic spectrum disorders or other pervasive developmental disorder.
* Has a history or clinical manifestations of significant metabolic (including diabetes mellitus, hypercholesterolemia, or dyslipidemia), hematologic, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urologic, immunologic, musculoskeletal, or psychiatric disorder unless currently controlled and stable with protocol-allowed medication for at least 30 days prior to Screening (except for ADHD in the age group of 6 to 11 years).
* Has sleep schedule changes required by employment, school and/or extra curricular activity (eg, shift worker) within 3 months prior to Screening, or has flown across greater than 3 time zones within 7 days prior to Screening.
* Has a history or clinical manifestations of depression, seizures, sleep apnea, restless leg syndrome, or periodic leg movements during sleep.
* Has a history of abdominal surgery (except laparoscopic cholecystectomy or uncomplicated appendectomy) or thoracic or nonperipheral vascular surgery within 6 months prior to study Day 1.
* Has a history of cancer, other than basal cell carcinoma or Stage 1 squamous cell carcinoma of the skin that has not been in remission for at least 5 years prior to study Day 1.
* Has used any tobacco (ie, nicotine) products (including but not limited to cigarettes, pipe, cigar, chewing tobacco, nicotine patch, or nicotine gum) within 6 weeks prior to Screening, or is unwilling to abstain from these products for the duration of the study.
* Has poor peripheral venous access.
* Has any clinically important abnormal finding as determined by a medical history, physical examination, electrocardiography (ECG), or clinical laboratory tests, as determined by the investigator. Participants with clinically significant abnormalities being considered for the study must be approved by both Takeda medical monitor or designee and the Principal Investigator.
* Has any additional condition(s) that in the Investigator's opinion would: a) affect sleep/wake function, b) prohibit from completing the study, or c) not be in the best interest of to participate in the study.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (2):
- United States (2):
  - Overland Park, Kansas
  - Kalamazoo, Michigan

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at one investigative site in the United States from 02 November 2009 to 03 April 2011.
Pre-assignment Details: Participants were enrolled into one of five treatment groups by age and assigned to either 4 mg or 8 mg ramelteon.
Groups:
- Children Ramelteon 4 mg: Children 6 to 11 years of age who had insomnia associated with Attention Deficit Hyperactivity Disorder (ADHD) received a single 4 mg oral dose of ramelteon.
Period: Overall Study
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Started | 6 | 6 | 8 | 8 | 28
Completed | 6 | 6 | 8 | 8 | 28
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg | Total
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28 | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 7.8 (1.72) | 9.2 (1.47) | 15.8 (1.67) | 15.5 (1.93) | 30.9 (10.17) | 21.7 (12.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 5 | 4 | 13 | 26
  Male | 3 | 5 | 3 | 4 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 5 | 7 | 8 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 0 | 0 | 5 | 9
  White | 1 | 5 | 8 | 8 | 23 | 45
  Multiracial | 2 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 8 | 8 | 28 | 56
Weight [Mean (Standard Deviation); unit: kg] | 28.1 (7.40) | 36.6 (12.24) | 61.4 (11.14) | 66.4 (12.99) | 76.8 (13.85) | 63.6 (21.40)
Height [Mean (Standard Deviation); unit: cm] | 128 (11.8) | 141 (11.9) | 168 (11.2) | 170 (12.8) | 174 (11.7) | 164 (19.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 16.5 (2.19) | 17.6 (3.75) | 21.7 (2.53) | 22.9 (2.94) | 25.1 (3.05) | 22.6 (4.29)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Maximum observed serum concentration (Cmax) is the peak serum concentration of ramelteon and its metabolite (M-II) after administration, obtained directly from the serum concentration-time curve.
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: The Pharmacokinetic (PK) set, which consisted of all patients who received study drug and had sufficient concentration data to calculate at least 1 PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
ng/mL
  Ramelteon (n=6, n=6, n=8, n=8, n=28) | 0.702 (0.8145) | 0.998 (1.0106) | 0.413 (0.4310) | 0.759 (0.5112) | 1.681 (2.3822)
  M-II (n=6, n=6, n=8, n=8, n=28) | 52.5 (21.83) | 79.0 (56.94) | 21.5 (6.54) | 39.6 (7.63) | 40.8 (14.53)

2. Primary Outcome: Time to Reach Maximum Serum Concentration (Tmax)
Description: Tmax: Time to reach the maximum serum concentration (Cmax) of ramelteon and its metabolite M-II, equal to time (hours) to Cmax.
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Median (Full Range); unit: hours
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
hours
  Ramelteon (n=6, n=6, n=7, n=8, n=28) | 0.50 [0.50 to 2.00] | 0.50 [0.50 to 2.00] | 2.00 [0.50 to 3.00] | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 3.00]
  M-II (n=6, n=6, n=8, n=8, n=28) | 0.75 [0.50 to 2.00] | 1.00 [0.50 to 2.00] | 2.00 [1.00 to 8.00] | 2.00 [0.50 to 2.00] | 2.00 [0.50 to 4.00]

3. Primary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc])
Description: Area under the serum concentration-time curve from time 0 to time of last quantifiable concentration (tlqc) of ramelteon and its metabolite M-II, calculated using the linear trapezoidal rule.
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
ng*hr/mL
  Ramelteon (n=6, n=6, n=8, n=8, n=28) | 0.703 (0.7098) | 1.353 (1.0621) | 1.022 (0.9553) | 1.564 (1.0591) | 3.636 (3.9104)
  M-II (n=6, n=6, n=8, n=8, n=28) | 127.2 (57.81) | 223.4 (61.84) | 88.8 (41.43) | 175.4 (43.39) | 190.6 (62.95)

4. Primary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUC[0-inf])
Description: Area under the serum concentration-time curve from time zero extrapolated to infinity for ramelteon and its metabolite M-II. The terminal area from the last quantifiable concentration (lqc) to infinity is calculated by approximation: lqc / terminal elimination rate constant (λz).
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 7 | 8 | 28
ng*hr/mL
  Ramelteon (n=4, n=5, n=4, n=8, n=25) | 1.03 (0.740) | 1.65 (1.104) | 1.75 (0.812) | 1.69 (1.051) | 4.22 (3.986)
  M-II (n=6, n=6, n=8, n=8, n=28) | 131.0 (59.67) | 227.6 (62.57) | 92.4 (43.68) | 179.2 (43.81) | 195.4 (65.06)

5. Primary Outcome: Apparent Clearance After Oral Administration (CL/F)
Description: Apparent oral clearance of drug from the serum calculated as:
  CL/F = Dose / Area under the serum concentration-time curve from time 0 extrapolated to infinity (AUC[0-inf]).
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 4 | 5 | 4 | 8 | 25
L/hr | 5374 (3117.6) | 6883 (4112.3) | 2605 (931.5) | 7319 (5426.6) | 4086 (3793.6)

6. Primary Outcome: Terminal Elimination Rate Constant (λz)
Description: The rate at which ramelteon and its metabolite M-II are eliminated from the body, calculated as the negative of the slope of the log-linear regression of the natural logarithm concentration-time curve during the terminal phase.
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
1/hour
  Ramelteon (n=4, n=5, n=4, n=8, n=25) | 0.743 (0.2181) | 0.659 (0.07205) | 0.550 (0.1358) | 0.541 (0.1651) | 0.483 (0.1234)
  M-II (n=6, n=6, n=8, n=8, n=28) | 0.436 (0.1109) | 0.363 (0.0771) | 0.377 (0.1217) | 0.331 (0.0936) | 0.278 (0.0400)

7. Primary Outcome: Terminal Elimination Half-life (T1/2)
Description: Terminal phase elimination half-life (T1/2) for ramelteon and its metabolite M-II is the time required for half of the drug to be eliminated from the serum, calculated as T1/2 = natural logarithm of 2 (ln[2]) / Terminal elimination rate constant (λz).
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
hours
  Ramelteon (n=4, n=5, n=4, n=8, n=25) | 1.02 (0.399) | 1.06 (0.117) | 1.32 (0.343) | 1.41 (0.490) | 1.52 (0.341)
  M-II (n=6, n=6, n=8, n=8, n=28) | 1.72 (0.635) | 1.98 (0.383) | 1.99 (0.536) | 2.21 (0.454) | 2.55 (0.385)

8. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Vz/F is the distribution of a drug between plasma and the rest of the body following oral administration, calculated as Vz/F = Apparent oral clearance (CL/F) / Terminal elimination rate constant (λz).
Time Frame: Day 1: predose (within 1 hour prior to dose) and at 0.5, 1, 2, 3, 4, 6, 8, 12, and 16 hours post-dose.
Population: Pharmacokinetic set where valid PK parameter estimates were available.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 4 | 5 | 4 | 8 | 25
Liters | 9136 (8703.1) | 10912 (6923.3) | 5016 (2462.4) | 14294 (10591.2) | 8606 (8417.1)

9. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product; it did not necessarily have to have a causal relationship with this treatment. The different categories of intensity (severity) were characterized as follows:
  Mild: The event was transient and easily tolerated by the participant.
  Moderate: The event causes the participant discomfort and interrupted usual activities.
  Severe: The event causes considerable interference with the participant's usual activities.
Time Frame: Day 1 to Day 15
Population: The safety set includes all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
participants
  Any AE | 0 | 1 | 1 | 0 | 3
  Mild AE | 0 | 1 | 1 | 0 | 2
  Moderate AE | 0 | 0 | 0 | 0 | 1
  Severe AE | 0 | 0 | 0 | 0 | 0
  Leading to discontinuation | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: Laboratory samples were collected at Screening, Check-in (Day 1), and Day 2 or Early Termination for assessment of hematology, chemistry, and urinalysis.
Time Frame: Screening, Day 1, Day 2 and Day 4
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
participants | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs included oral body temperature, pulse and blood pressure (taken after 5 minutes in the sitting position). Vital signs measurements were determined to be clinically significant according to predefined criteria.
Time Frame: Screening, Day 1, Day 2 and Day 4
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
participants | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram Findings
Description: A standard 12-lead electrocardiogram (ECG) was recorded at Screening, Day 2, and at Final Visit (Day 4). The investigator interpreted the ECG using one of the following categories: within normal limits, abnormal but not clinically significant, or abnormal and clinically significant.
Time Frame: Screening, Day 2 and Day 4
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
participants | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Physical Examination Results
Description: A complete physical examination was performed for each participant at Screening, Check-in (Day 1), Day 2, and Final Visit (Day 4) or Early Termination. The examination consisted of a review of the following body systems: eyes; ears, nose, and throat; respiratory; gastrointestinal; extremities; musculoskeletal; cardiovascular; nervous; and dermatological.
Time Frame: Screening, Day 1, Day 2 and Day 4
Population: Safety set.
Measure: Number; unit: participants
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Number analyzed (Participants) | 6 | 6 | 8 | 8 | 28
participants | 0 | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 15.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Children Ramelteon 4 mg | Children Ramelteon 8 mg | Adolescents Ramelteon 4 mg | Adolescents Ramelteon 8 mg | Healthy Adult Ramelteon 8 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/8 | 0/28
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 1/8 | 0/8 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Children Ramelteon 4 mg (N=6) | Children Ramelteon 8 mg (N=6) | Adolescents Ramelteon 4 mg (N=8) | Adolescents Ramelteon 8 mg (N=8) | Healthy Adult Ramelteon 8 mg (N=28)
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights therefrom or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.